CLINICAL TRIAL: NCT01117337
Title: Comparing Non-fixation of Mesh to Mesh Fixation in Laparoscopic Total Extraperitoneal Inguinal Hernia Repair Under Spinal Anesthesia- A Randomized Controlled Trial
Brief Title: Comparing Non-fixation of Mesh to Mesh Fixation in Laparoscopic Inguinal Hernia Repair
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Moulana Hospital (Other)
Responsible Party: Mohamed Ismail, Moulana Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MH-ECN-04-08
Record Dates: First submitted 2010-05-03; First posted 2010-05-05 (Estimated); Results first posted 2010-08-31 (Estimated); Last update posted 2010-08-31 (Estimated); Status verified 2008-07

CONDITIONS: Inguinal Hernia
Keywords: Hernia, laparoscopic, recurrence, pain, inguinal
MeSH Terms: conditions — Hernia, Inguinal; Hernia; Recurrence; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mesh Non Fixation Group (No Intervention): Laparoscopic Total extraperitoneal repair of Inguinal hernia under Spinal Anesthesia - Mesh is not fixed by ant means
  Interventions: Procedure: Mesh Fixation

INTERVENTIONS:
Procedure: Mesh Fixation — Laparoscopic Total extraperitoneal repair of Inguinal hernia under Spinal Anesthesia - Mesh is not fixed to any structure
  Other Names: Mesh fixation by Tacker

SUMMARY:
The purpose of the study is

1. To compare the recurrence rate of the laparoscopic total extra peritoneal inguinal hernia repair without fixation of the mesh to mesh fixation under spinal anesthesia
2. To test whether non-fixation of mesh leads to less pain compared to the repair when the mesh is fixed.

DETAILED DESCRIPTION:
Hernia repair is one of the most common surgery performed all over the world. The same is true about India. With more than a billion population, the number of hernia patients in India perhaps run in millions. The laparoscopic repair is increasingly becoming popular in India.

Decreased post operative pain and lesser morbidity are the main advantages of Total Extra Peritoneal Repair (TEP) over open hernia repair. Laparoscopic hernia repair is now recommended as the method of choice for bilateral and recurrent inguinal hernias. The disadvantages of TEP are requirement of general anesthesia (GA), need to fix the mesh, seroma formation and difficult learning curve. Fixation of mesh with metal staples, apart from increasing the cost, may lead to new post operative groin pain which even becomes chronic in small percentage of patients. This had led to various studies showing that the non-fixation of mesh is safe, cost effective and lead to no increased risk of hernia recurrence compared to the conventional open hernia repair. Requirement of GA for TEP repair also had several disadvantages compared to regional anesthesia such as significant hemodynamic changes, delayed recovery, post operative nausea and vomiting, increased cost and inability to give anesthesia in high cardio-pulmonary risk patients. Several studies in recent past have demonstrated TEP is feasible and safe in regional anesthesia (epidural or spinal) as well. We earlier reported that TEP repair could be done without fixation of the mesh under regional anesthesia.

This study is a Randomized Controlled Trial (RCT) comparing the outcome of non-fixation of mesh during laparoscopic inguinal hernia repair with fixation of mesh under spinal anesthesia. The end points measured would be the recurrence of the hernia and pain in the post operative period.

ELIGIBILITY:
Inclusion Criteria:

* All reducible inguinal hernias will be included in the study

Exclusion Criteria:

* Irreducible hernia after anesthesia
* Obstructed and strangulated hernias
* Pediatric hernias
* Associated other hernias like ventral hernias
* Unfit for spinal anesthesia

Ages: 16 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2008-09; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Ismail, MBBS, MS, Principal Investigator — Moulana Hospital
Locations (1):
- Moulana Hospital, Perintalmanna, Kerala, India

REFERENCES:
- [Background] Garg P, Rajagopal M, Varghese V, Ismail M. Laparoscopic total extraperitoneal inguinal hernia repair with nonfixation of the mesh for 1,692 hernias. Surg Endosc. 2009 Jun;23(6):1241-5. doi: 10.1007/s00464-008-0137-0. Epub 2008 Sep 24. PMID 18813990
- [Background] Taylor C, Layani L, Liew V, Ghusn M, Crampton N, White S. Laparoscopic inguinal hernia repair without mesh fixation, early results of a large randomised clinical trial. Surg Endosc. 2008 Mar;22(3):757-62. doi: 10.1007/s00464-007-9510-7. Epub 2007 Sep 21. PMID 17885789
- [Background] Ferzli GS, Frezza EE, Pecoraro AM Jr, Ahern KD. Prospective randomized study of stapled versus unstapled mesh in a laparoscopic preperitoneal inguinal hernia repair. J Am Coll Surg. 1999 May;188(5):461-5. doi: 10.1016/s1072-7515(99)00039-3. PMID 10235572
- [Derived] Garg P, Nair S, Shereef M, Thakur JD, Nain N, Menon GR, Ismail M. Mesh fixation compared to nonfixation in total extraperitoneal inguinal hernia repair: a randomized controlled trial in a rural center in India. Surg Endosc. 2011 Oct;25(10):3300-6. doi: 10.1007/s00464-011-1708-z. Epub 2011 May 2. PMID 21533969

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between September to December 2008, 120 patients with inguinal hernia presented to randomization at Moulana Hospital, Perianthalmanna, Kerala, India.
Pre-assignment Details: 15 patients didn't meet inclusion criteria and one patient didn't give consent. 104 patients were randomized to mesh fixation (52 patients) and mesh non-fixation (52 patients). One month and one year follow-up was completed in 100 patients. The follow-up ranged from 15-19 months with a median of 16.2 months.
Groups:
- Mesh Fixation Group: Laparoscopic Total extraperitoneal repair of Inguinal hernia under Spinal Anesthesia - Mesh is fixed with two tackers
- Mesh Non Fixation Group: The patients in whom the mesh was not fixed by any means
Period: Overall Study
Arm/Group | Mesh Fixation Group | Mesh Non Fixation Group
Started | 52 (52 pateints on inguinal hernia were randomized to mesh fixation group) | 52
Underwent Surgery | 52 (52 patients underwent surgery) | 52
Completed | 48 (48 completed one year follow-up. 4 lost to follow-up.) | 52
Not Completed | 4 | 0
Not completed — Lost to Follow-up | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mesh Fixation Group | Mesh Non Fixation Group | Total
Number analyzed (Participants) | 52 | 52 | 104
Age Continuous [Mean (Standard Deviation); unit: years] | 47.2 (12.9) | 51.9 (16.8) | 49.6 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 51 | 49 | 100

OUTCOME MEASURES:

1. Primary Outcome: Recurrence of Inguinal Hernia on the Operated Side in Mesh Non-fixation and Mesh Fixation Group.
Description: Patients in both the arms will be followed up post operatively at 24 hours, 1 week, 1 month and 1 year to check for recurrence or persistence of inguinal hernia on the operated side. At these follow up visits, the patients would be asked about reoccurence of bulge on the operated side and will be examined clinically. In case, there is a suspicion of recurrence, the patient would be examined by a second surgeon and undergo Ultrasound and/or CT to confirm the recurrence of hernia.
Time Frame: 1 year
Measure: Number; unit: Participant
Arm/Group | Mesh Fixation Group | Mesh Non Fixation Group
Number analyzed (Participants) | 48 | 52
Participant | 0 | 0

2. Primary Outcome: Proportion of Patients Having Pain in the Post Operative Period
Description: To compare the proportion of patients having pain in the mesh fixation and non fixation group at one month postoperatively.
Time Frame: 1 month
Measure: Number; unit: Participant
Arm/Group | Mesh Fixation Group | Mesh Non Fixation Group
Number analyzed (Participants) | 48 | 52
Participant | 3 | 8
Statistical Analysis 1: Comparison: Mesh Fixation Group vs Mesh Non Fixation Group; Test type: Superiority or Other; p = 0.2, Fisher Exact

3. Secondary Outcome: Seroma Formation
Description: A seroma was defined as a non tender, irreducible hemispherical swelling with a fluctuant or firm consistency at the hernia site, examined and found during the first year. The diagnosis was based on the clinical finding of a palpable fluid collection without a size limit. One could get above the upper border of the swelling and there was usually absence of a cough impulse. To detect seroma, the clinical examination was carried at the first follow-up visit on the 7th postoperative day.
Time Frame: One year
Measure: Number; unit: Participant
Arm/Group | Mesh Fixation Group | Mesh Non Fixation Group
Number analyzed (Participants) | 48 | 52
Participant | 5 | 8
Statistical Analysis 1: Comparison: Mesh Fixation Group vs Mesh Non Fixation Group; Test type: Superiority or Other; p = 0.56, Fisher Exact

ADVERSE EVENTS:
Arm/Group | Mesh Fixation Group | Mesh Non Fixation Group
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/52
Other Adverse Events (participants affected / at risk) | 0/48 | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No